CLINICAL TRIAL: NCT00521209
Title: Improving Health Habits: Self-Care Priorities
Brief Title: Patient-Directed Lifestyle Change and Health Promotion Program or Usual Care in Low-Income, Uninsured Participants in Los Angeles County, California
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-002325; R21CA112441-01 (NIH); UCLA-G-060801501A; CDR0000561559 (Other: UCLA)
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2023-08-08 (Actual); Status verified 2023-05

CONDITIONS: Impoverished Population
Keywords: Impoverished Population

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinic 1 - intervention (Experimental): Clinic 1 will feature the Self-Care Stimulating Disease Prevention Program (SCSDPP) intervention
  Interventions: Behavioral: Self-Care Stimulating Disease Prevention Program (SCSDPP)
- Clinic 2 - no intervention (Other): Clinic 2 will continue with standard procedures no intervention
  Interventions: Other: Stand procedures, no intervention

INTERVENTIONS:
Behavioral: Self-Care Stimulating Disease Prevention Program (SCSDPP) — The SCSDPP development is guided by the following premises: a) patient-directed lifestyle change or "self-prescription" of behavior change is potentially a more empowering, sustainable, and proactive approach to addressing personal health habits than the more conventional physician-directed approach; b) patient-directed lifestyle change or "self-prescription" of behavior change is potentially an important predictor of self-efficacy and long-term adherence to healthy habits; c) behavior change in isolation is less sustainable than change that is reinforced by other distinct but related changes (e.g., the potential synergy of improving diet and physical activity concurrently to prevent chronic disease); d) a multi-level change directed at the service delivery system and physician support, however small, has the added benefit of potentially reducing provider and staff burden while maximizing available clinic and community resources; and f) brief physician counseling
  Arms: Clinic 1 - intervention
Other: Stand procedures, no intervention
  Arms: Clinic 2 - no intervention

SUMMARY:
RATIONALE: Clinic-based health programs may be effective in improving the diets and physical activity levels of low-income, uninsured participants in Los Angeles County, California.

PURPOSE: This randomized clinical trial is studying a patient-directed lifestyle change and health promotion program to see how well it works compared with usual care in low-income, uninsured participants in Los Angeles County, California.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the feasibility and impact of a clinic-based intervention protocol in Los Angeles county, California, for improving the dietary choices and physical activity levels of low-income clinic populations in Los Angeles County, California.

OUTLINE: The two participating clinics are randomly assigned to provide care as outlined below to participants who routinely visit that clinic.

* Arm I (clinic 1, intervention program): Physicians provide health advice to the participants for 1-2 minutes using a motivational interviewing technique during a regularly scheduled appointment. Health messages to motivate changes in diet and physical activity levels are tailored to the participant based on information from the Patient Health Behavior Priority Assessment (PHBPA). Physicians also create a mutually agreed upon self-directed lifestyle change plan (the Health Priority Plan) for the participant using information from the PHBPA. Participants undergo a 10-minute interview to indicate whether the doctor discussed the plan and their satisfaction with the visit. After the first clinic encounter, participants are contacted by a health educator via telephone 4 times over a 2-month period. The telephone sessions are designed to identify obstacles and challenges in adhering to the Health Priority Plan and help participants to persevere with the plan. Participants are followed at baseline, 2 months, and 6 or 12 months. Participants have blood pressure and weight measured and blood collected to determine levels of nutrients and fat and sugar content during these follow-up visits.
* Arm II (clinic 2, control program): Physicians provide usual care during a regularly scheduled appointment. Participants are followed at baseline, 2 months, and 12 months. Participants have blood pressure and weight measured and a subset of participants also have blood collected to determine levels of nutrients and fat and sugar content during these follow-up visits.

In both arms, participants also undergo a 30-minute interview about diet and physical activity and take a step test to measure heart rate and oxygen level during the follow-up visits. All participants undergo an exit interview at the end of the study about their perceptions of the program and what can be improved in the study. Participants' medical record information is examined for the period of 12 months prior to enrollment in the study, during the 12-month study period, and for 12 months after the exit interview date.

PROJECTED ACCRUAL: A total of 140 participants (40 for arm I and 100 for arm II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Receiving care at one of two study sites within the Venice Family Clinic network of clinics: Simms-Mann Clinic or Rose Avenue Clinic

  * Must remain in the Los Angeles area during the 12-month study period
* Low income level and uninsured, and therefore at increased risk for nutrition- and lifestyle-related health conditions, including overweight, obesity, and cancer
* Shows interest in changing diet and physical activity behavior as indicated by response to Patient Health Behavior Priority Assessment (PHBPA)
* No history of cancer, except non-melanoma skin cancer or in situ cancers
* Prticipated in the focus group discussion or cognitive interview for the pre-intervention portion of the study (IRB #G06-08-014-01)

PATIENT CHARACTERISTICS:

* English- or Spanish-speaking
* Accessible by telephone where they can be contacted over time during the study to conduct follow-up health education phone calls
* Willing to cooperate with data collection (e.g., lab draws, completing interviews, etc.)
* Not pregnant
* No medical condition precluding free choice of foods (e.g., colitis, irritable bowel syndrome, or diabetes)
* No medical condition precluding participation in common forms of aerobic or resistance exercise, including any of the following:

  * Uncontrolled angina
  * Severe asthma or hypertension
  * Severe physical impairment that requires a wheelchair, cane, or special bed
  * Congestive heart failure
  * Nephropathy from any cause
  * Chronic pulmonary disease
* No cognitive impairment

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects that have behavior changes as a result of using the Self-Care Stimulating Disease Prevention Program | Through study completion, expected to be 10 years

SECONDARY OUTCOMES:
Ease of integration of the SCSDPP into the community health clinic setting through the number of subjects that implement life style changes | Through study completion, expected to be 10 years

CONTACTS AND LOCATIONS:
Overall Officials: William McCarthy, PhD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No